CLINICAL TRIAL: NCT05556746
Title: A Phase IIc, Open-Label, Randomized Controlled Trial of Ultra-Short Course Bedaquiline, Clofazimine, Pyrazinamide and Delamanid Versus Standard Therapy for Drug-Susceptible Tuberculosis (PRESCIENT)
Brief Title: Ultra-Short Course Bedaquiline, Clofazimine, Pyrazinamide and Delamanid Versus Standard Therapy for Drug-Susceptible TB
Acronym: PRESCIENT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Cape Town (Other); Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other); University of Stellenbosch (Other); University of California, Los Angeles (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Serena Patricia Koenig, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022p003075; U01AI170426 (NIH)
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Tuberculosis, Pulmonary; HIV
Keywords: Pulmonary Tuberculosis; Treatment Shortening; HIV; Drug-Susceptible Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — bedaquiline; Clofazimine; Pyrazinamide; OPC-67683; Rifampin; Isoniazid; Ethambutol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to the experimental or standard groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCZD (Experimental): Bedaquiline 200 mg for 12 weeks + pyrazinamide 1000 - 2000 mg (according to weight) for 12 weeks + clofazimine 300 mg for 2 weeks, followed by 100 mg for 10 weeks + delamanid 200 mg for 12 weeks, all given once daily.
  Interventions: Drug: Bedaquiline; Drug: Clofazimine; Drug: Pyrazinamide; Drug: Delamanid
- Standard TB Treatment (Active Comparator): Rifampin, isoniazid, ethambutol and pyrazinamide for 8 weeks, followed by rifampin and isoniazid for 18 weeks; given daily in fixed dose combinations at standard weight-based doses.
  Interventions: Drug: Rifampin; Drug: Isoniazid; Drug: Ethambutol; Drug: Pyrazinamide

INTERVENTIONS:
Drug: Bedaquiline — Daily therapy for 12 weeks
  Arms: BCZD
Drug: Clofazimine — Daily therapy for 12 weeks
  Arms: BCZD
Drug: Pyrazinamide — Daily therapy for 12 weeks
  Arms: BCZD
Drug: Delamanid — Daily therapy for 12 weeks
  Arms: BCZD
Drug: Rifampin — Daily therapy for 26 weeks
  Arms: Standard TB Treatment
Drug: Isoniazid — Daily therapy for 26 weeks
  Arms: Standard TB Treatment
Drug: Ethambutol — Daily therapy for 8 weeks
  Arms: Standard TB Treatment
Drug: Pyrazinamide — Daily therapy for 8 weeks
  Arms: Standard TB Treatment

SUMMARY:
The PRESCIENT trial is a Phase IIc, open-label, randomized trial that will compare a 12-week regimen of bedaquiline (BDQ), clofazimine (CFZ), pyrazinamide (PZA), and delamanid (DLM) with standard treatment for drug-susceptible pulmonary tuberculosis. Eligible participants will be randomized in a 1:1 ratio to BDQ, CFZ, PZA, and DLM (BCZD) or standard anti-TB therapy.

Participants in the experimental arm with evidence of poor clinical response at the end of therapy will be re-treated with standard TB therapy. The primary analysis is a superiority efficacy comparison of time to liquid culture conversion through 8 weeks in the experimental (BCZD) arm vs. the standard therapy arm. The other key secondary outcome is safety.

DETAILED DESCRIPTION:
The PRESCIENT trial is a Phase IIc, open-label, randomized trial that will compare a 12-week regimen of bedaquiline (BDQ), clofazimine (CFZ), pyrazinamide (PZA), and delamanid (DLM) with standard treatment for drug-susceptible pulmonary tuberculosis. Eligible participants will be randomized in a 1:1 ratio to BDQ, CFZ, PZA, and DLM (BCZD) or standard anti-TB therapy. Randomization will be stratified by presence of lung cavitation and HIV status.

Participants will be randomized to one of two arms:

Arm 1 (Experimental): BDQ 200 mg for 12 weeks + PZA 1000 - 2000 mg (according to weight) for 12 weeks + CFZ 300 mg for 2 weeks, followed by 100 mg for 10 weeks + DLM 200 mg for 12 weeks, all given once daily.

Arm 2 (Standard of Care): RIF, INH, EMB and PZA for 8 weeks, followed by RIF and INH for 18 weeks.

Medications will be given daily in fixed dose combinations at standard weight-based doses. Adherence will be supported through automated reminders and monitored remotely in real time with Wisepill electronic adherence monitoring devices or with directly observed treatment. Participants in the experimental arm with evidence of poor clinical response will be re-treated with standard TB therapy. The primary analysis is a superiority efficacy comparison of time to liquid culture conversion through 8 weeks in the experimental (BCZD) arm vs. the standard therapy arm. Participants will have extended post-treatment follow up to evaluate clinical efficacy as a secondary composite outcome measure at 86 weeks after randomization (74 weeks after completion of experimental therapy, when most relapses are expected to occur). The other key secondary outcome is safety, measured as the proportion with new Grade 3 or higher adverse events; we shall focus on QTcF prolongation and hepatitis as adverse events of special interest. Through an efficient Phase IIc design, the PRESCIENT trial will test microbiological efficacy, evaluate safety, and detect treatment-emergent resistance with the ultra-short BCZD regimen. PRESCIENT will provide rapid evidence for microbiological efficacy as well as key information on safety and clinical treatment outcomes to inform the feasibility and promise of a subsequent phase III treatment-shortening trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained and signed.
* Male or female, aged ≥18 years.
* Pulmonary TB diagnosed by Xpert MTB/RIF, Xpert MTB/RIF Ultra, Line Probe Assay (LPA), or mycobacterial culture.
* Sputum positive for acid fast bacilli (at least 1+ grade on the WHO scale).
* Pulmonary TB diagnosed without known INH resistance (by LPA or Xpert MTB/XDR) and without known RIF resistance (by either LPA or Xpert). Note that phenotypic DST for INH resistance will be done on screening cultures (using MGIT). If baseline molecular or phenotypic test results that become available after enrollment detect resistance to INH or RIF, the participant will be a late exclusion from the study.
* Newly diagnosed with TB and have a history of being untreated for at least 6 months after cure from a previous episode of TB.
* For participants living with HIV, CD4+ cell count ≥200 cells/mm3, obtained within 30 days prior to study entry. Enrollment of participants living with HIV will be limited to no more than 20% of the total study population.
* For participants living with HIV, must be currently receiving or planning to initiate ART at or before study week 8.
* Laboratory values at study screening:

  * Alanine aminotransferase (ALT) ≤3x the upper limit of normal (ULN)
  * Total bilirubin ≤2.5 x ULN
  * Creatinine ≤2 x ULN
  * Potassium ≥3.5 mEq/L, ≤5.5 mEq/L
  * Absolute neutrophil count (ANC) ≥650/mm3
  * Hemoglobin ≥7.0g/dL
  * Platelet count ≥50,000/mm3
* For females of reproductive potential, negative serum or urine pregnancy test within 5 days prior to entry and willingness to use effective contraception for the duration of the study. Female participants who are not of reproductive potential must have documentation of menopause, hysterectomy, or bilateral oophorectomy or bilateral tubal ligation. Acceptable forms of contraception include: condoms, intrauterine device or intrauterine system, cervical cap with spermicide, diaphragm with spermicide.
* The initial 25% of enrollment will be restricted to participants (n = 39) with mild or moderate disease, defined as having sputum with higher Xpert MTB/RIF cycle threshold (Ct) values (> 17 cycles) and the absence of extensive lung disease on chest X-ray (involvement of at least half of the area of the entire thoracic cavity). Thereafter, all eligible patients will be offered participation without a pause in enrollment.

Exclusion Criteria:

* More than 5 days of treatment directed against active TB for the current TB episode preceding study entry.
* Current extrapulmonary TB (e.g. neurological, skeletal, abdominal, or nodal), not including pleural TB, in the opinion of the site investigator.
* Pregnant or breastfeeding.
* Weight <30kg.
* Inability to take oral medications.
* Current or planned use of any drug known to severely prolong the QTc interval, including, but not limited to: amiodarone, amitriptyline, chloroquine, chlorpromazine, cisapride, disopyramide, erthyromycin, moxifloxacin, procainamide, quinidine, or sotalol.
* Current or planned use of one or more of the following HIV medications: HIV protease inhibitors, HIV non-nucleoside reverse transcriptase inhibitors, elvitegravir/cobicistat, or bictegravir.
* Current or past use of clofazimine, bedaquiline or delamanid.
* QTcF >450ms for men or >470 ms for women.
* Current or history of known personal or family long QT syndrome.
* Known allergy/sensitivity to components of study TB drugs or their formulation.

Microbiologic confirmation of drug-susceptible TB is not always available at the time of enrollment. Enrolled individuals who are subsequently determined to meet either of the following criteria will be classified as late exclusions and study treatment will be discontinued. These participants will be transitioned to routine care but requested to remain in study follow up for safety evaluations.

A. Screening, baseline study, and Week 1 visit sputum cultures fail to grow M. tuberculosis.

B. Resistance to RIF or INH is detected from baseline molecular or phenotypic testing results that become available after enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time to stable liquid culture conversion | Measured through Week 8
  Defined as the first of two negative sputum cultures, consecutive or not, without an intervening positive culture, and/or visits wherein the participant is unable to produce sputum and has no signs or symptoms of active TB.

SECONDARY OUTCOMES:
Proportion experiencing any Grade 3 or higher AE | Measured at Week 60
  AE includes any occurrence that is new in onset or aggravated at least one-grade from baseline.
  AE's will be graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, July 2017.
Proportion with favorable composite outcome | Measured at Week 60
  Defined as no failure, relapse, or non-accidental death
Proportion who prematurely discontinue treatment | Measured at Week 12 in experimental group and Week 26 in standard group
  Defined as discontinuation other than due to violent death, natural disaster, or administrative censoring
Change in skin coloration at weeks 8, 12, 16, 26, 60, and 86 | Measured through Week 86
  Mean change in subjective 10-point numeric rating scale where 0=none, 10=worst possible change in coloration
Distress related to skin coloration at weeks 8, 12, 16, 26, 60, and 86 | Measured through Week 86
  Mean subjective distress related to skin coloration on 10-point rating scale where 0=non, 10-worst possible distress due to coloration
Mean change in QTcF from baseline to week 1, 2, 4, 8, 12, and 16 | Measured through Week 16
  The QTcF is derived from ECG readings, which the sites conduct in triplicate (three ECGs 5-10 minutes apart). The mean of all measurements (up to 3) that are readable and available will be used at each of baseline (screening visit), Week 2, Week 8, Week 12, and Week 16.
Mean change in QTcF from baseline to end of treatment | Measured at Week 12 in Arm 1 and Week 26 in Arm 2
  The QTcF is derived from ECG readings, which the sites conduct in triplicate (three ECGs 5-10 minutes apart). The mean of all measurements (up to 3) that are readable and available will be used at baseline (screening visit), week 12 (Arm 1) and week 26 (Arm 2).
Occurrence of absolute QTcF ≥480 ms and <500 ms, and ≥500 ms | Measured through Week 16
  The QTcF is derived from ECG readings, which the sites conduct in triplicate (three ECGs 5-10 minutes apart). The mean of all measurements (up to 3) that are readable and available will be used at week 16 in Arm 1 and Arm 2
Occurrence of QTcF change from baseline of ≥30 ms and <60 ms, and ≥60 ms | Measured through Week 16
  The QTcF is derived from ECG readings, which the sites conduct in triplicate (three ECGs 5-10 minutes apart). The mean of all measurements (up to 3) that are readable and available will be used at week 16 in Arm 1 and Arm 2
Proportion of participants with one or more serious adverse events (SAEs) | Week 86
  Serious adverse events reported at any time during participation in the trial
Proportion with culture conversion in liquid and solid media (separately) at weeks 4, 8 and 12 after randomization | Measured at Weeks 4, 8, and 12
  Proportion of participants who have achieved stable culture conversion, defined as two negative sputum cultures, consecutive or not, without an intervening positive culture and/or visits wherein the participant is unable to produce sputum and has no signs of active TB; occurring before or at the week 4, 8, or 12 visit, respectively.
Proportion with TB relapse (by M. tuberculosis genotyping) from end of treatment to 86 weeks | Measured through Week 86
  For participants who had successful culture conversion through the end of study treatment, TB relapse is defined as a recurrence of TB emanating from the same strain as the participant's originally diagnosed TB, which will be determined through whole genome sequencing.
Proportion of treatment-emergent genotypic and phenotypic resistance to BCZD | Measured through Week 86
  For participants in experimental group only. MIC values will be evaluated against resistance-associated variants for paired baseline and failure isolates. Frequencies and proportions with phenotypic and/or genotypic resistance to any drug will be reported.
Time (days) to positivity in liquid culture (MGIT) after start of treatment across study arms | Measured through Week 8
  Median (Q1, Q3) times to positivity in liquid culture at each time point (Weeks 1, 2, 3, 4, 6, and 8) in Arm 1 and Arm 2.
Time to stable liquid culture conversion | Measured through Week 12
  Defined as the first of two negative sputum cultures, consecutive or not, without an intervening positive culture, and/or visits wherein the participant is unable to produce sputum and has no signs or symptoms of active TB

CONTACTS AND LOCATIONS:
Overall Officials: Serena Koenig, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Sean Wasserman, MBChB, PhD, Principal Investigator — University of Cape Town
Locations (2):
- GHESKIO, Port-au-Prince, Haiti
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Where possible, we will make raw data available in publications (directly or through online appendices). Although the final dataset will be stripped of identifiers prior to release for sharing, we believe there remains the possibility of deductive disclosure of subjects with unusual characteristics. We will therefore make the data and associated documentation available to users under a controlled access process/data-sharing agreement, in compliance with current international standards to protect participant confidentiality.
  Where applicable, data documentation and de-identified data will be deposited for sharing along with demographics consistent with applicable laws and regulations. Data content, format, and organization will conform with relevant data and terminology standards.
Supporting Information: Study Protocol, SAP, ICF